CLINICAL TRIAL: NCT04632407
Title: Can Flaxseed Prevent Broken Hearts in Women With Breast Cancer Study?
Acronym: CANFLAX
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Boniface Hospital (Other)
Responsible Party: Principal Investigator, Dr. Davinder S. Jassal, Professor of Medicine, St. Boniface Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CT/2019/CANFLAX
Record Dates: First submitted 2020-10-21; First posted 2020-11-17 (Actual); Last update posted 2020-11-17 (Actual); Status verified 2020-11

CONDITIONS: Cardiotoxicity
Keywords: Cardiotoxicity; Chemotherapy; Flaxseed
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Intervention Model Description: The study participants will be randomized to either oat fibre "milk" or flax "milk"
Who Masked: Participant, Care Provider, Investigator
Masking Description: The 2 products (oat fibre "milk" and flax "milk") are assigned a unique ID code.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flax "milk" (Experimental): A total of 30 women will receive flax (FLX) "milk" on a daily basis for a total of 4 months. The FLX "milk" will be composed of BevPur (30 mesh FLX), various gums for texture, vanilla flavoring, several minor ingredients, and water. Each serving contains 15 grams of FLX and 3.75 grams of Omega-3.
  Interventions: Dietary Supplement: Flax "milk"
- Oat fibre "milk" (Experimental): A total of 30 women will receive the oat fiber "milk" on a daily basis for a total of 4 months. The oat fibre "milk" will be composed of oat fibre, various gums for texture, vanilla flavoring, several minor ingredients, and water.
  Interventions: Dietary Supplement: Oat fibre "milk"

INTERVENTIONS:
Dietary Supplement: Flax "milk" — See above
  Arms: Flax "milk"
Dietary Supplement: Oat fibre "milk" — See above
  Arms: Oat fibre "milk"

SUMMARY:
The main goal of the current research program is to examine the use of nutraceuticals, in particular flaxseed (FLX), in the prevention of Doxorubicin and Trastuzumab (DOX+TRZ) mediated cardiotoxicity in the clinical setting. As Manitoba continues to be one of the top FLX producers in the world, there is an increasing public awareness of the importance of the consumption of this whole grain commodity in the prevention of cancer and cardiovascular disease. In North America, approximately 1 in 8 women will develop breast cancer and will receive treatment with DOX+TRZ. Although women with breast cancer are at risk of developing heart failure due to chemotherapy, FLX has the capacity to prevent this outcome. The purpose of the CANFLAX study is to establish FLX "milk" as an effective method in preventing heart failure in women with breast cancer.

DETAILED DESCRIPTION:
Cardiovascular toxicity is a potential short and long-term complication of anti-cancer therapy with DOX+TRZ in the breast cancer setting. Although FLX is commonly consumed in up to 30% of women with breast cancer to improve overall disease burden and survival, it is important to study whether this natural dietary agent can also reduce the cardiotoxic side effects of DOX+TRZ in the clinical setting. The investigators hypothesize that the prophylactic consumption of FLX "milk" will prevent adverse cardiovascular remodeling and improve overall functional capacity in women with breast cancer receiving DOX+TRZ therapy. The two specific aims of the CANFLAX study include: Aim 1: FLX "milk" will prevent the development of heart failure in women with early stage breast cancer (EBC) who are treated with DOX+TRZ based chemotherapy; and Aim 2: FLX "milk" will improve cardiac functional capacity in this patient population.

ELIGIBILITY:
Inclusion Criteria:

* i) ≥18 years old;
* ii) women with newly diagnosed early stage breast cancer (Stage I-IIIA)
* iii) chemotherapy with 5 fluorouracil, epirubicin, and cyclophosphamide (FEC) or adriamycin and cyclophosphamide (AC) for 4 months

Exclusion Criteria:

* i) pre-existing diagnosis of heart failure and/or LVEF<40%
* ii) pre-existing use of anti-hypertensive agents including ACE inhibitors (ACEi) or beta blockers
* iii) planned use of any herbal/antioxidant/fatty acid/nutritional supplements at any time in the duration of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) change | 1 year
  Left ventricular ejection fraction (LVEF %) will be evaluated using transthoracic echocardiography at baseline and 12 month follow-up. A difference in LVEF>10% from baseline will be considered significant.

CONTACTS AND LOCATIONS:
Overall Officials: Davinder S Jassal, MD, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface Albrechtsen Research Centre, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No